CLINICAL TRIAL: NCT01436383
Title: Oxidative Stress in Hypobaric Hypoxia and Influence on Vessel-tone Modifying Mediators
Brief Title: Oxidative Stress in Hypobaric Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Kantonsspital Aarau (Other)
Responsible Party: Prof. Dr. med. A. R. Huber, Center of Laboratory Medicine, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK 1189; SNSF 3200B0-108300
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Hypobaric Hypoxia; Metabolomics; Oxidative Stress; Acute Mountain Sickness
Keywords: high altitude; hypobaric hypoxia; metabolomics; oxidative stress; acute mountain sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Hypoxic exposure — Hypoxic exposure

SUMMARY:
The trial investigates changes in metabolism during high altitude expedition up to 6865m. A mass-spectrometry based platform is used to detect different oxidative stress related metabolites. Symptoms of acute mountain sickness are evaluated and correlated with laboratory parameters.

DETAILED DESCRIPTION:
Background

Altitude related illness, which include acute mountain sickness (AMS), high altitude pulmonary edema (HAPE) and high altitude cerebral edema (HACE), is common in subjects exposed to high altitude during professional or leisure time activities. There are independent risk factors such as: individual susceptibility and rate of ascent. HAPE is a potentially life-threatening complication of high altitude stay, mostly occuring within the first 2-5 days of exposure. Although there is a controversial discussion, excessive hypoxic pulmonary vasoconstriction is thought to be the main trigger for developing HAPE. Beside the controversial discussion if hypobaric hypoxia leads to oxidative stress it is not known whether oxidative stress contributes to AMS or HAPE.

Objective

The investigators hypothesize that reactive oxygen species are generated during high altitude stay and contribute to the development of acute mountain sickness. Furthermore they would like to describe other changes in metabolic pathways possibly contributing to vessel tone dysregulation.

Methods

36 healthy volunteers will examined during an high altitude medical research expedition to Mount Muztagh ata (7549m) in Western China. Acute mountain sickness scores and clinical parameters will be assessed. Metabolomics analysis of more than 390 parameters, using a mass spectrometry-based targeted metabolomic platform, is used to detect systemic oxidative stress and functional impairment of enzymes that require oxidation-sensitive co-factors. Furthermore routine laboratory test will be done, for example CRP, creatinine and interleukines

ELIGIBILITY:
Inclusion Criteria:

* healthy
* physical fit
* mountaineering experience
* 18-70 years

Exclusion Criteria

* any type of disease
* regular intake of medicaments
* history of high altitude pulmonary edema
* severe acute mountain sickness below an altitude of 3500m
* any history of high altitude cerebral edema

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of volunteers with acute mountain sickness | during ascent, expected to be approximately 19-23 days

SECONDARY OUTCOMES:
Change from baseline in oxygen saturation in blood | during ascent, expected to be approximately 19-23 days
Changes from baseline in oxidative stress | during ascent, expected to be approximately 19-23 days
Changes from baseline in different metabolic pathways | during ascent, expected to be approximately 19-23 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Huber, Prof. Dr. med., Study Chair — Center of Laboratory Medicine, Cantonal Hospital Aarau, 5001 Aarau
Locations (1):
- Center of Laboratory Medicine, Aarau, Switzerland